CLINICAL TRIAL: NCT06458478
Title: Effects of the Application of a Hyper-oxygenated Gel After Extraction of Impacted Lower Third Molars: Randomized Controlled Study
Brief Title: Effects of the Application of a Hyper-oxygenated Gel After Oral Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera di Perugia (Other)
Responsible Party: Principal Investigator, Mitro Valeria, Principal Investigator, Azienda Ospedaliera di Perugia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMF2
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Molar, Fourth; Extracting Own Teeth; Edema Face; Pain; Trismus
Keywords: dysodontiasis; third molar; oral surgery; edema; trismus; pain
MeSH Terms: conditions — Tooth, Supernumerary; Pain; Trismus; Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyper-oxygenated Gel (Active Comparator): Patients undergoing lower third molar extraction. Post-operatively, the antibiotic (amoxicillin + clavulanic acid) and the painkiller (paracetamol 1000mg x 2 times a day x 7 days) are prescribed.
  Furthermore, patients will have to use the Novox drop at the post-extraction site 3 times a day for 7 days (without taking liquids for 30 minutes after use).
  Interventions: Other: Hyper-oxygenated gel
- Placebo (Placebo Comparator): Patients undergoing lower third molar extraction. Post-operatively, the antibiotic (amoxicillin + clavulanic acid) and the painkiller (paracetamol 1000 mg x 2 times a day x 7 days) are prescribed.
  Furthermore, patients will have to use the Placebo, glycerin based gel, at the post-extraction site 3 times a day for 7 days (without taking liquids for 30 minutes after use).
  Interventions: Other: glycerin based gel

INTERVENTIONS:
Other: Hyper-oxygenated gel — Novox drop is a medical device (CE certified, class II b, non-invasive) based on oxygen-enriched olive oil (Excipients: Mint essential oil (2%), Stevia extract (1%)). Mechanism of action: facilitate the healing process by creating, thanks to the release of reactive oxygen species (ROS), a microenvironment favorable to the activation of the microcirculation and at the same time unfavorable to the proliferation of pathogens. Furthermore, it has a film-forming, protective, barrier and soothing action thanks to its oily nature.
  Other Names: Novox drop
  Arms: Hyper-oxygenated Gel
Other: glycerin based gel — The placebo consists of a viscous, colorless and transparent gel, based on glycerin (Conformity:FUI).
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate whether the topical application of Novox® Drop on surgical wounds after the extraction of lower third molars can have a clinical advantage.

The primary objective of the study is to evaluate the possible reduction of masseteric trismus (masticatory muscle spasm - primary outcome) and of post-operative pain and facial edema (swelling - secondary outcomes) after the extraction of impacted third molars compared to those who do not use it (placebo=glycerin-based gel).

DETAILED DESCRIPTION:
Novox drop is a medical device (CE certified, class II b, non-invasive) based on oxygen-enriched olive oil (Excipients: Mint essential oil (2%), Stevia extract (1%)). Mechanism of action: facilitate the healing process by creating, thanks to the release of reactive oxygen species (ROS), a microenvironment favorable to the activation of the microcirculation and at the same time unfavorable to the proliferation of pathogens. Furthermore, it has a film-forming, protective, barrier and soothing action thanks to its oily nature.

The placebo consists of a viscous, colorless and transparent gel, based on glycerin (Conformity:FUI).

The company producing Novox Drop will package both gels in opaque disposable syringes, identical from each other and distinguishable only by the presence of an "A" or "B" code. During the phases of the study, only the company will be aware which of the two codes will be associated with the medical device and which will be associated with the placebo. The patients to be subjected to the study will be obtained from those arriving at the maxillofacial surgery clinics for the surgical extraction of complex lower third molars, starting from July 2024 until the necessary sample size of 72 participants is reached. Each of them, who will be assigned a sequential numerical code, will be placed randomly (randomized) in one of the two arms of the study itself, group A or group B, using the Excel Microsoft 2015 system.

Patients in group A, in addition to the standard antibiotic therapy (amoxicillin + clavulanic acid 1 g x 3 times a day x 7 days) and painkiller (paracetamol 1000 mg x 2 times a day x 7 days) will be prescribed the home use of syringe A. Patients in group B, in addition to the aforementioned traditional therapy, the syringe B. The gel prescribed in both groups must be applied to the post-extraction site 3 times a day for 7 days. Furthermore, after each application of the gels, the patient cannot consume drinks and solid foods for 30 minutes.

The duration of the study will be one week, and will be divided into three visits:

the first at time 0 as soon as the surgery is finished where all the hygiene recommendations will be made, the basic therapy drugs (antibiotic and anti-inflammatory) will be prescribed, and the gels will be prescribed in the A or B syringes; the second visit at time 1 three days after the operation and the third visit at time 2 after a week in which the patient's health status will be assessed, the study data will be collected, the blisters of the therapy performed will be collected and the hygiene advice will be reiterated .

For the administration method just described, the study will be a triple blind study, where neither the patient, nor the prescribing doctor nor the observer of the results of the surgical wounds will be aware of the type of gel used. Only the doctor responsible for cataloging and processing complete with the results you will be aware of which gel was contained in syringe A and which in syringe B.

ELIGIBILITY:
Inclusion Criteria:

* good systemic and local health conditions of the patient;
* age between 18 and 35 years;
* understanding of the Italian language,
* indications for the extraction of impacted bilateral lower third molars (38 and 48) according to the criteria reported in the classifications of Winter and that of Pell and Gregory;
* the root of the impacted third molars is completely formed.

Exclusion Criteria:

* diabetes mellitus;
* systemic arterial hypertension;
* hyperthyroidism;
* osteoporosis;
* immunosuppressed;
* osteonecrosis of the jaws;
* pregnancy;
* patients with mandibular third molars in position C according to "the Pell & Gregory Classification" on the radiological measurements (angles and positions) for which third molar extraction surgery is required.;
* local alterations such as pericoronitis, odontogenic cysts and tumors in relation to the third molars;
* allergies;
* ordinary use of analgesics or antibiotics by the patient.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Masseteric trismus. | seven days
  Masseteric trismus will be assessed by measuring the width of the mouth opening. Precisely, the distance in cm between the mesial corners of the incisal edges of the upper central incisors and the lower right incisors at maximum mouth opening, before surgery and on the seventh postoperative day, using a caliper. Measurements will be taken twice to determine the average score. The difference between the average of each postoperative measurement and the preoperative one will indicate the trismus for that day.

SECONDARY OUTCOMES:
Post-operative pain | seven days
  The intensity of postoperative pain will be assessed with a Visual Analog Scale (VAS). The patient will be able to express the degree of pain perceived at both time one and time two on a scale of ten intervals. Grade 1 on the scale indicates no pain, grade ten indicates very intense pain.
Facial swelling | seven days
  The swelling of the face in cm will be determined by measuring the distance from the corner of the mouth to the attachment of the earlobe following the curvature of the cheek and the distance from the outer canthus of the eye to the corner of the jaw. The arithmetic mean of the two measurements will be considered as reference. The difference between each postoperative measurement and baseline will indicate facial swelling for that day.

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Gilli, Dr, Principal Investigator — Azienda Ospedaliera Perugia
Locations (1):
- Ospedale Santa Maria della Misericordia, Perugia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim HS, Noh SU, Han YW, Kim KM, Kang H, Kim HO, Park YM. Therapeutic effects of topical application of ozone on acute cutaneous wound healing. J Korean Med Sci. 2009 Jun;24(3):368-74. doi: 10.3346/jkms.2009.24.3.368. Epub 2009 Jun 12. PMID 19543419
- [Background] Valacchi G, Fortino V, Bocci V. The dual action of ozone on the skin. Br J Dermatol. 2005 Dec;153(6):1096-100. doi: 10.1111/j.1365-2133.2005.06939.x. PMID 16307642
- [Background] Bocci V. Biological and clinical effects of ozone. Has ozone therapy a future in medicine? Br J Biomed Sci. 1999;56(4):270-9. PMID 10795372
- [Background] Martinez-Sanchez G, Al-Dalain SM, Menendez S, Re L, Giuliani A, Candelario-Jalil E, Alvarez H, Fernandez-Montequin JI, Leon OS. Therapeutic efficacy of ozone in patients with diabetic foot. Eur J Pharmacol. 2005 Oct 31;523(1-3):151-61. doi: 10.1016/j.ejphar.2005.08.020. Epub 2005 Sep 29. PMID 16198334
- [Background] Montevecchi M, Dorigo A, Cricca M, Checchi L. Comparison of the antibacterial activity of an ozonated oil with chlorhexidine digluconate and povidone-iodine. A disk diffusion test. New Microbiol. 2013 Jul;36(3):289-302. Epub 2013 Jun 30. PMID 23912871
- [Background] Osunde OD, Saheeb BD. Effect of age, sex and level of surgical difficulty on inflammatory complications after third molar surgery. J Maxillofac Oral Surg. 2015 Mar;14(1):7-12. doi: 10.1007/s12663-013-0586-4. Epub 2013 Oct 1. PMID 25729220
- [Background] Amin MM, Laskin DM. Prophylactic use of indomethacin for prevention of postsurgical complications after removal of impacted third molars. Oral Surg Oral Med Oral Pathol. 1983 May;55(5):448-51. doi: 10.1016/0030-4220(83)90227-x. PMID 6575332
- [Background] Marques RV, Branco-de-Almeida LS, Marques DM, Oliveira IC, Mendes SJ, Rodrigues VP, Lopes FF. Effect of the intra-alveolar administration of dexamethasone on swelling, trismus, and pain after impacted lower third molar extraction: a randomized, double-blind clinical trial. Med Oral Patol Oral Cir Bucal. 2022 Jan 1;27(1):e51-e58. doi: 10.4317/medoral.24894. PMID 34564685
- [Background] Cinquini C, Marchionni S, Derchi G, Miccoli M, Gabriele M, Barone A. Non-impacted tooth extractions and antibiotic treatment: A RCT study. Oral Dis. 2021 May;27(4):1042-1051. doi: 10.1111/odi.13607. Epub 2020 Sep 4. PMID 32790913
- [Background] Olmedo-Gaya MV, Manzano-Moreno FJ, Munoz-Lopez JL, Vallecillo-Capilla MF, Reyes-Botella C. Double-blind, randomized controlled clinical trial on analgesic efficacy of local anesthetics articaine and bupivacaine after impacted third molar extraction. Clin Oral Investig. 2018 Dec;22(9):2981-2988. doi: 10.1007/s00784-018-2386-1. Epub 2018 Feb 15. PMID 29450738
- [Background] Hadad H, Santos AFP, de Jesus LK, Poli PP, Mariano RC, Theodoro LH, Maiorana C, Souza FA. Photobiomodulation Therapy Improves Postoperative Pain and Edema in Third Molar Surgeries: A Randomized, Comparative, Double-Blind, and Prospective Clinical Trial. J Oral Maxillofac Surg. 2022 Jan;80(1):37.e1-37.e12. doi: 10.1016/j.joms.2021.08.267. Epub 2021 Sep 6. PMID 34656515